CLINICAL TRIAL: NCT04114877
Title: Perinatal Attentional Retraining Intervention for Smoking (PARIS) for Minority Women
Brief Title: Perinatal Attentional Retraining Intervention for Smoking for Minority Women
Acronym: PARIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1008007245; 1R21MD012697-01A1 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Smoking Relapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- attentional retraining (AR) (Experimental): Cognitive bias modification (CBM) procedures are interventions aimed at changing the impulsive (automatic) processes that underlie unhealthy behaviors such as smoking. Attentional retraining (AR) is the most commonly used CBM intervention in the study of addiction-related attentional bias.
  Interventions: Behavioral: Attentional retraining (AR)
- visual probe (VP) (Active Comparator): The visual probe (VP) task can measure attentional bias for drug-related cues.
  Interventions: Behavioral: Visual probe (VP)

INTERVENTIONS:
Behavioral: Attentional retraining (AR) — Cognitive bias modification (CBM) procedures are interventions aimed at changing the impulsive (automatic) processes that underlie unhealthy behaviors such as smoking. AR is the most commonly used CBM intervention in the study of addiction-related attentional bias. The idea behind AR is to reduce attentional bias and therefore minimize exposure to drug cues, because attention to such stimuli may provoke craving and undermine cessation attempts.
  Arms: attentional retraining (AR)
Behavioral: Visual probe (VP) — The visual probe (VP) task can measure attentional bias for drug-related cues. In the typical VP task, a pair of pictures or words (e.g. one smoking-related and one neutral) is briefly presented simultaneously side by side on a computer screen. After the pictures disappear, a probe stimulus (e.g. a small dot) is presented in the location that had been occupied by one of the pictures (or words), and participants are required to press a key as quickly as possible in response to the probe. Attentional bias for drug-related cues is detected by a faster response to a probe that replaces a drug-related stimulus (vs. a neutral stimulus), since attention will have been preferentially allocated to that area of visual display. The traditional VP task only assesses attentional bias, and does not modify it in any way.
  Arms: visual probe (VP)

SUMMARY:
The proposed research intends to randomize 50 abstinent pregnant Black or Hispanic smokers to receive either the attentional retraining (AR) or control VP task. Participants will be asked to carry around a smartphone as they go about their daily lives for 2 weeks in their last month of pregnancy (Phase 1).

The smartphone will sound an alert randomly during the day, at which time participants will be asked to respond to a short set of questions assessing subjective states; this will be followed by a request to complete the AR (or control) procedures. This same procedure will be repeated for 2 weeks immediately after delivery (Phase 2).

Women will undergo a follow-up visit 3 months after the end of Phase 2, and complete an unmodified VP and follow-up assessments.

DETAILED DESCRIPTION:
There are 2 specific aims that this study intends to address.

Specific Aim 1: To examine whether AR delivered on a smartphone can modify attentional bias to smoking-related stimuli and craving for tobacco cigarettes.

Specific Aim 2: To examine whether AR delivered on a smartphone can modify attentional bias to stress-related stimuli and reduce perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of smoking 5+ cigarettes per day that have achieved abstinence during pregnancy by 32 weeks gestation.
* The ability to speak and write English.
* An Edinburgh Postnatal Depression Scale (EPDS) score <10.

Exclusion Criteria:

* Current substance abuse (e.g., alcohol, benzodiazepines, marijuana).
* Current major depressive disorder, minor depression or dysthymia, or history of any of these disorders in the last 6 months.
* The presence of an Axis I psychotic disorder.
* Plans to relocate out of the area.
* Imminent incarceration.
* Planned inpatient hospitalization during study period.
* Plans to breastfeed. Women who plan to breastfeed will be excluded since this is a powerful, independent motivation for remaining abstinent and may decrease the relapse event rate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna Forray, MD, Principal Investigator — Associate Professor of Psychiatry; Psychiatry Director, Adult Sickle Cell Program; Co-Director, Center for Wellbeing of Women and Mothers
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP) | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Customized [Count of Participants; unit: Participants]
  >30 years | 10 | 4 | 14
  ≤30 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic, White | 2 | 1 | 3
  Hispanic, Black | 3 | 1 | 4
  Black, non-Hispanic | 8 | 6 | 14
  >1 Race, non-Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22
Education [Count of Participants; unit: Participants]
  < High school degree | 1 | 2 | 3
  High school degree | 5 | 2 | 7
  Some college (no degree) | 5 | 5 | 10
  Associate's degree | 1 | 0 | 1
  Refuse to Answer | 1 | 0 | 1
Pre-quit smoking level [Count of Participants; unit: Participants]
  ≤10 cigarettes/day | 11 | 5 | 16
  >10 cigarettes/day | 2 | 4 | 6
Anxiety [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 9 | 4 | 13
Age started smoking (years) [Mean (Standard Deviation); unit: years] | 15.8 (3.2) | 15.9 (1.5) | 15.8 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Attentional Bias- Smoking Related Stimuli
Description: Attentional bias (AB) is assessed using the standard (unmodified) visual probe (VP) task on the smartphone and study visits, and measured by the reaction time (RT) in milliseconds, i.e. the time it takes a participant to identify the location of the probe after presentation of the stimulus. The AB scores will be computed as the difference in RTs on trials where the probe replaced the smoking picture vs. trials where the probe replaced the neutral picture. The VP task can measure attentional bias for drug-related cues. In the typical VP task, a pair of pictures or words (e.g. one smoking-related and one neutral) is briefly presented simultaneously side by side on a computer screen. After the pictures disappear, a probe stimulus (e.g. a small dot) is presented in the location that had been occupied by one of the pictures (or words), and participants are required to press a key as quickly as possible in response to the probe.
Time Frame: end of phase 2, up to 3 months
Population: While 13 participants were randomized to AR and 9 to the control VP task, only 10 and 4 participants, respectively, provided sufficient data to be included in the analysis.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
Number analyzed (Participants) | 10 | 4
milliseconds | -44.0 (170.9) | 37.9 (163.6)
Statistical Analysis 1: Comparison: Attentional Retraining (AR) vs Visual Probe (VP); Test type: Superiority; p > 0.05, Mixed Models Analysis; Linear mixed models

2. Primary Outcome: Attentional Bias Toward Stressrelated Stimuli
Description: Attentional bias (AB) is assessed using the standard (unmodified) visual probe (VP) task on the smartphone and at study visits, and measured by the reaction time (RT) in milliseconds, i.e. the time it takes a participant to identify the location of the probe after presentation of the stimulus. The AB scores will be computed as the difference in RTs on trials where the probe replaced the stress-related word vs. trials where the probe replaced the neutral word. The VP task can measure attentional bias for drug-related cues. In the typical VP task, a pair of pictures or words (e.g. one smoking-related and one neutral) is briefly presented simultaneously side by side on a computer screen. After the pictures disappear, a probe stimulus (e.g. a small dot) is presented in the location that had been occupied by one of the pictures (or words), and participants are required to press a key as quickly as possible in response to the probe.
Time Frame: end of phase 2, up to 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
Number analyzed (Participants) | 10 | 4
milliseconds | -12.1 (130.6) | -46.5 (94.8)
Statistical Analysis 1: Comparison: Attentional Retraining (AR) vs Visual Probe (VP); Test type: Superiority; p > 0.05, Mixed Models Analysis; Linear mixed models

3. Secondary Outcome: Self-reported Craving
Description: Self-reported craving is a single item used to assesses craving for cigarettes ("I have strong urges to smoke a cigarette") on a 7-point Likert scale (1 = Strongly Disagree, 7 = Strongly Agree) in the daily assessments delivered on the smartphone and at study visits. Higher scores on the 7-point Likert scale are indicative of higher cravings for cigarettes, with a 7 indicating high craving for a cigarette and 1 indicating low craving for a cigarette. This scale is a subjective measure of a participant's craving for cigarettes developed by the researchers and utilized in prior research.
Time Frame: end of phase 2, up to 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on 7-point Likert scale
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
Number analyzed (Participants) | 10 | 4
score on 7-point Likert scale | 1.35 (0.89) | 1.66 (1.82)
Statistical Analysis 1: Comparison: Attentional Retraining (AR) vs Visual Probe (VP); Test type: Superiority; p > 0.05, Mixed Models Analysis; Linear mixed models

4. Secondary Outcome: Self-reported Stress
Description: Self-reported stress was assessed using four items: three adapted from the Parenting Stress Index (I feel I can't handle things; I feel trapped by parenting; I feel overwhelmed by trying to meet my baby's needs) and one item developed for the study (since the last assessment my baby has been difficult to console). Participants responded to the four items on 7-point Likert-type scales (1 = Strongly Disagree, 7 = Strongly Agree) in the daily assessments delivered on the smartphone and at study visits. The mean score was computed. Higher scores on the scale are indicative of high stress levels and low scores of low stress levels.
Time Frame: end of phase 2, up to 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
Number analyzed (Participants) | 10 | 4
score on a scale | 3.34 (0.77) | 3.57 (0.70)
Statistical Analysis 1: Comparison: Attentional Retraining (AR) vs Visual Probe (VP); Test type: Superiority; p > 0.05, Mixed Models Analysis; Linear mixed models

5. Secondary Outcome: Smoking Relapse
Description: Relapse is defined as any smoking on 7 consecutive days or smoking at least once each week over 2 consecutive weeks. Smoking history is collected with the timeline follow-back at each study visit. This is a binary yes/no outcome. Presented here is the number of participants who relapsed to smoking.
Time Frame: from randomization to 6-month follow-up, up to 8 months
Population: While 13 participants were randomized to AR and 9 to the control VP task, only 8 and 4 participants, respectively, provided sufficient data to be included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
Number analyzed (Participants) | 8 | 4
Participants | 4 | 2
Statistical Analysis 1: Comparison: Attentional Retraining (AR) vs Visual Probe (VP); Test type: Superiority; p = 0.455, Fisher Exact

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Attentional Retraining (AR) | Visual Probe (VP)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 0/13 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04114877/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04114877/ICF_000.pdf